CLINICAL TRIAL: NCT04164160
Title: Effectiveness of the Integrated Care Model Salut+Social in Patients With Chronic Conditions: a Mixed Methods Study Protocol
Brief Title: An Integrated Care Model for Chronic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 7Z18/020
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2019-10

CONDITIONS: Integrated Care
Keywords: Integrated care; Health and social care; Chronic disease; Primary Health Care; Quality of life
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- integrated-care-model benefiting group (Experimental): Chronic patients whose clinical and social data will be added in the integrated care model application software.
  Interventions: Other: integrated-care-model benefiting group

INTERVENTIONS:
Other: integrated-care-model benefiting group — Patients will be called for the ﬁrst interview of the study by the healthcare professional. Their data will be automatically entered in the Salut + Social app, they will be asked to respond to the study questionnaires (ad hoc questionnaire for sociodemographic data, EuroQol-5D, Zarit questionnaire and Morisky-Green test) and will take part in the future actions to be planned for them. Patients will receive an appointment to attend their PCC at 6, 9, and 12 months after their incorporation into the program. In those follow-up, the same questionnaires will be provided together with the IEXPAC questionnaire, which evaluates the experience of the chronic patient with the new care model.

SUMMARY:
Integrated care models aim to promote the coordination and communication between services. The present study aim to evaluate the effectiveness of a new integrated care model (Salut+Social model) which will promote the coordination and communication between social and healthcare services in southern Catalonia (Spain) for the improvement of quality of life of chronic patients, adherence to treatment, access to medical services and caregiver overload. Also, we will evaluate the experience of health and social professionals with the new model implemented.

DETAILED DESCRIPTION:
A clinical trial with mixed methodology will be carried out. The intervention consists of the promotion and coordination between the social and health sectors, for 6 months, through the use of information and communication technology (ICT) tools that operate as an interface for the integrated care model. The study subjects are chronic patients with health and social conditions that are susceptible to be treated in a collaborative and coordinated way in the field of primary health care. A sample size of 141 patients was estimated. Questionnaires will be used at baseline and at 6, 9 and 12 months after the beginning of the study for the evaluation of quality of life, treatment adherence, medical service and caregiver overload. The principal variable is the quality of life. For statistical analysis, comparisons of means and proportions at different time points will be performed. One discussion group will be performed with the aim of improving the care model according to professionals' opinions. A thematic content analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with at least one health and one social condition, as below specified:

  1. health condition, according to diagnosis of the electronic medical history: complex chronic patient; advanced chronic disease; patient in the home care program; dementia; neurodegenerative diseases; stroke; others chronic disease.
  2. social condition, according to social service workstation from Ribera d'Ebre district: dependence grade; home social service assistance; teleassistance systems assigned by home support.
* Knowledgement of Spanish or Catalan.
* Accepting participation in the study (with informed consent signed by the patient or by the caregiver).

Exclusion Criteria:

* Institutionalized patients.
* Users with difficulties filling out or respond a questionnaire.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in life quality | change from life quality at 6, 9 and 12 months after the beginning of the study.
  to be evaluated with the EuroQol- 5 Dimension (EQ-5D). It will be measured by a scale Likert: 0 (worst) to 1 (best).
Change in caregiver burden | change from Zarit Caregiver Burden Inventory at 6, 9 and 12 months after the beginning of the study.
  to be evaluated with the Zarit Caregiver Burden Inventory. It will be measured by a scale Likert: 22 (best) to 110 (worst).
Change in adherence to treatment | change from Morisky and Green test at 6, 9 and 12 months after the beginning of the study.
  be evaluated with the Morisky and Green test. It will be measured with a dichotomic variable: compliant (if response for the 4 questions is: No/Yes/No/No); noncompliant (if response for the 4 questions is different for: No/Yes/No/No).
Change in patient experience about his/her care | change from IEXPAC at 6, 9 and 12 months after the beginning of the study
  Be evaluated with the IEXPAC (Instrument for the Evaluation of the Chronic Patient's Experience). Each of the 11 items will be measured with 5-point Likert scale. The global punctuation is an average of the score of the each of the items: 0 (worst experience) to 10 (best experience).

SECONDARY OUTCOMES:
Sociodemographic characteristics of the patients | baseline (pre intervention period)
  age, sex, level of education, civil status, job situation, nationality
Caregiver characteristics: caregiver with family relationship | baseline (pre intervention period)
  To be evaluated with an ad hoc questionnaire (yes/no type)
Caregiver characteristics: caregiver relationship | baseline (pre intervention period)
  To be evaluated with an ad hoc questionnaire (1. Couple; 2. Mother; 3. Father; 4. Son; 5. Others).
Caregiver characteristics: hours of support | baseline (pre intervention period)
  To be evaluated with an ad hoc questionnaire (quantitative variable).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català de la Salut, Tortosa, Tarragona, Spain

REFERENCES:
- [Derived] Gavalda-Espelta E, Del Mar Lleixa-Fortuno M, Baucells-Lluis J, Ferre-Ferrate M, Mora-Lopez G, Tomas-Navarro B, Curto-Romeu C, Lucas-Noll J, Aguilar Martin C, Goncalves AQ, Ferre-Grau C. Effectiveness of the integrated care model Salut+Social in patients with chronic conditions: A mixed methods study protocol. Medicine (Baltimore). 2020 May;99(19):e19994. doi: 10.1097/MD.0000000000019994. PMID 32384454